CLINICAL TRIAL: NCT03656835
Title: A Pilot Study of Nanochip Technology for Monitoring Treatment Response and Detection of Relapse in Patients With Diffuse Large B-Cell Lymphoma
Brief Title: Nanochip Technology in Monitoring Treatment Response and Detecting Relapse in Participants With Diffuse Large B-Cell Lymphoma
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Responsible Party: Principal Investigator, Beth Christian, Principal Investigator, Ohio State University Comprehensive Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: OSU-18154; NCI-2018-01536 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2018-08-30; First posted 2018-09-04 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Diffuse Large B-Cell Lymphoma; Diffuse Large B-Cell Lymphoma Germinal Center B-Cell Type; Diffuse Large B-Cell Lymphoma, Not Otherwise Specified; High Grade B-Cell Lymphoma
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Diagnostic (ILN biochip testing) (Experimental): Participants' blood samples undergo ILN biochip testing at diagnosis, before and after every course of chemotherapy, every 3 months for 2 years, and at relapse.
  Interventions: Procedure: Molecular Nanotechnology

INTERVENTIONS:
Procedure: Molecular Nanotechnology — Undergo ILN biochip testing
  Other Names: MNT

SUMMARY:
This trial studies how well nanochip technology (immuno-tethered lipoplex nanoparticle [ILN] biochip) works in monitoring treatment response and in detecting relapse in participants with diffuse large B-cell lymphoma. Finding genetic markers for diffuse large B-cell lymphoma may help identify participants with this disease and help predict the outcome of treatment. It is not yet known how well ILN biochip-based testing monitors treatment response or detects relapse in participants with diffuse large B-cell lymphoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine whether ILN biochip can be used to detect molecular marker(s) to monitor treatment response in patients with newly diagnosed diffuse large B-cell lymphoma (DLBCL).

II. Determine whether ILN biochip can promote early detection of disease relapse in patients with DLBCL.

OUTLINE:

Participants' blood samples undergo ILN biochip testing at diagnosis, before and after every course of chemotherapy, every 3 months for 2 years, and at relapse.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed treatment naive DLBCL. Subtypes including high grade B-cell lymphoma, not otherwise specified (NOS) and de-novo DLBCL including germinal center B-cell type (GCB) and non-GCB subtypes.
* Intent to receive entire care (treatment and follow-up) at Ohio State University (OSU).
* Receiving treatment with curative intent.
* Receiving planned 6 cycles of chemotherapy.
* Ability to consent.

Exclusion Criteria:

* Transformed lymphomas.
* DLBCL with leukemic presentation.
* Primary central nervous system (CNS) lymphoma.
* Participating in other clinical trial/ receiving experimental therapy.
* Patients with a "currently active" second malignancy that, in the opinion of the principal investigator, will interfere with patient participation, or confound data interpretation.
* Pregnancy (positive serum or urine pregnancy test) or breast feeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2018-09-26 (Actual); Primary Completion 2024-11-20 (Actual); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Treatment response | Up to 2 years
  The association of the expression measured by immuno-tethered lipoplex nanoparticle (ILN) biochip and quantitative reverse transcription polymerase chain reaction (qRT-PCR) will be displayed by scatter plot. Receiver operating characteristic (ROC) curves and corresponding area under the curves (AUCs) will be calculated and compared. With these data collected serially over time, patterns will be explored graphically using trace plots showing the trend across treatment for each individual participant.
Early detection of relapse | Up to 2 years
  Changes in expression between baseline and relapse will be summarized with descriptive statistics and explored graphically.

CONTACTS AND LOCATIONS:
Overall Officials: Beth Christian, MD, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (1):
- Ohio State University Comprehensive Cancer Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The Jamesline — http://cancer.osu.edu